CLINICAL TRIAL: NCT04771975
Title: Connecting Breast Cancer Survivors for Exercise: A Randomized Controlled Trial Phase I and II
Brief Title: Connecting Breast Cancer Survivors for Exercise
Acronym: C4E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jenna Smith (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor-Investigator, Jenna Smith, Post Doctoral Fellow (Catherine Sabiston PI), University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: I2I1
Record Dates: First submitted 2020-02-28; First posted 2021-02-25 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: exercise; physical activity; oncology; breast cancer; survivorship; social support; resistance training; body image; physical self; body functionality
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MatchQEP group (Experimental): Phase 1: All participants will receive an 'Exercise Peer Support Guide' that provides suggestions for supporting their exercise partner and a one-page document describing current exercise guidelines for cancer survivors [16-18]. All participants will also be given a Fitbit device, which will be used for device-measured MVPA.
  Participants in the MatchQEP group will receive exercise information and program sessions tailored by a qualified exercise professional (QEP) specifically for each BCS in the dyad. Dyads will meet with the QEP via Zoom once per week for 10 weeks for up to 60 minutes. For four weeks following the 10-week intervention period, the QEP will be available for consultation (i.e., a post-intervention tapering period) as needed by the MatchQEP group participants.
  Phase 2: Was not an RCT (i.e., all Phase 1 participants were approached to participate in Phase 2). Phase 2 is a pre-post intervention design, with no control group.
  Interventions: Behavioral: Exercise Counselling; Behavioral: Partner Matching; Behavioral: Resistance training sessions led by a QEP
- Match group (Active Comparator): Phase 1: All participants will receive an 'Exercise Peer Support Guide' that provides suggestions for supporting their exercise partner and a one-page document describing current exercise guidelines for cancer survivors [16-18]. All participants will also be given a Fitbit device, which will be used for device-measured MVPA.
  Participants in the Match (control) group will independently communicate and support each other around exercise for 10 weeks. They will not have any contact with a QEP during this time.
  Phase 2: Was not an RCT (i.e., all Phase 1 participants were approached to participate in Phase 2). Phase 2 is a pre-post intervention design, with no control group.
  Interventions: Behavioral: Partner Matching; Behavioral: Resistance training sessions led by a QEP

INTERVENTIONS:
Behavioral: Exercise Counselling — Phase 1: See previous description for MatchQEP (Intervention) group. Phase 2: Was not an RCT (i.e., all Phase 1 participants were approached to participate in Phase 2). Phase 2 is a pre-post intervention design, with no control group. Phase 2 participants had the option to extend their time in the study for an additional 8-weeks, which includes an online virtual (zoom) resistance training program with a qualified exercise professional (QEP) with a new study partner. The 8-week program was open to all participants from Phase 1 who choose to continue in the study, regardless of initial randomization status. Behavioural and exercise counselling were offered to phase 2 participants.
  Other Names: QEP support
  Arms: MatchQEP group
Behavioral: Partner Matching — Phase 1: All participants will be matched with another participant (fellow BCS) and will facilitate / support exercise with their partner for the duration of the study.
  Phase 2: Was not an RCT (i.e., all Phase 1 participants were approached to participate in Phase 2). Phase 2 is a pre-post intervention design, with no control group. Phase 2 participants were rematched with different partner for this phase of the trial.
  Participants will be matched based on personal and cancer-related characteristics.
Behavioral: Resistance training sessions led by a QEP — Phase 2: participants were offered the option to extend their time in the study for an additional 8-weeks, which includes an online virtual (zoom) resistance training program with a qualified exercise professional (QEP) with a new study partner.

SUMMARY:
Phase 1: The purpose of this study is to examine interpersonal and individual effects of partnering BCS with a peer and a qualified exercise professional (QEP) on self-reported exercise volume (MVPA; primary outcome), and device-measured exercise volume (MVPA; Fitbit), social support, and HRQOL (secondary outcomes). Cost-effectiveness and intervention adherence will also be explored as tertiary outcomes. The effects of a peer and QEP-support intervention group, labelled MatchQEP, will be compared to a control group of BCS who are matched with a peer, but not a QEP, labelled Match.

Phase 2: The purpose of this study is to examine whether the addition of 8-weekly QEP-lead resistance training Zoom sessions with an exercise partner interacts with social support (i.e., tangible, informational, emotional) and how this interaction relates to overall exercise volume as an extension of Phase 1 (one year after phase 1 was completed). A secondary aim of Phase 2 is to examine the direct influence of resistance training on body image, self-efficacy, the physical self, and body functionality among the participants.

DETAILED DESCRIPTION:
The purpose of this project is to examine naturally occurring social support as related to daily exercise behavior. In our ecological momentary assessment (EMA) study, the function of social support (tangible, informational, emotional) was be explored as independent variables, and exercise dose (minutes, intensity) and type (aerobic, resistance training, flexibility) will be examined as dependent variables. The associations will be used to inform motivational and behaviour change messaging in ActiveMatch, a program developed and run by the PI of this study, Dr. Catherine Sabiston. It is generally hypothesized that the provision of social support will be associated with greater exercise behaviour. In phase 1 of Connect for exercise, the RCT portion of this study, the addition of qualified exercise professional (QEP) support will be evaluated compared to social support from a participant match (exercise partner) alone. In Phase 2 of the Connect for exercise trial (pre-post design with no control group), we will examine whether the addition of 8-weekly QEP-lead resistance training Zoom sessions with an exercise partner interacts with social support (i.e., tangible, informational, emotional) and how this interaction relates to overall exercise volume (completed one-year post phase 1 completion). A secondary aim of Phase 2 is to examine the direct influence of resistance training on body image, self-efficacy, the physical self, and body functionality among the participants. There is evidence that resistance training improves these outcomes in women (Santa Barbara et al., 2017), but the relationship is understudied in breast cancer survivors. Improvements in these outcomes have, in turn, been related to increases in PA and sustainable positive PA outcomes. Considering the decreases in body image and body functionality appreciation reported by BCS during and after treatment (Resaei et al., 2016), this relationship warrants further investigation.

ELIGIBILITY:
Phase 1 and phase 2:

Inclusion Criteria:

* Female
* Breast cancer survivors
* Stage 1-4 cancer
* Aged >18 years
* Have been cleared for exercise
* Have consistent access to an Internet-connected device
* Currently exercise ≤ 150 minutes per week.

Exclusion Criteria:

* Report contraindications to exercise such as physical disability
* Had recent or planned reconstructive surgery
* Have no consistent access to an Internet-connected device
* Are currently meeting exercise guidelines (performing > 150 minutes of moderate-to- vigorous exercise)
* Have not been cleared to participate in exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Phase 1 and Phase 2: Change in exercise volume | Baseline, 10-weeks post baseline.
  The Godin Leisure Time Exercise Questionnaire will be used to measure exercise volume over 1 week. It is a self-report measure which asks respondents to give weekly frequencies and durations of strenuous, moderate, and mild aerobic activities and resistance training sessions. Together responses are summed to determine a total weekly leisure activity score. It is shown to be reliable and valid (r=.53) when classifying respondents into 'insufficiently active' and 'active' categories (Amireault & Godin, 2015; Amireault et al., 2015; Amireault et al., 2015; Godin & Shephard, 1985b). Respondents are classified as 'active' by exceeding a score of 24 on this scale (Amireault & Godin, 2015; Amireault et al., 2015; Amireault et al., 2015).
Phase 1 and Phase 2: Change in exercise volume | 14-weeks post baseline
  The Godin Leisure Time Exercise Questionnaire will be used to measure exercise volume over 1 week. It is a self-report measure which asks respondents to give weekly frequencies and durations of strenuous, moderate, and mild aerobic activities and resistance training sessions. Together responses are summed to determine a total weekly leisure activity score. It is shown to be reliable and valid (r=.53) when classifying respondents into 'insufficiently active' and 'active' categories (Amireault & Godin, 2015; Amireault et al., 2015; Amireault et al., 2015; Godin & Shephard, 1985b). Respondents are classified as 'active' by exceeding a score of 24 on this scale (Amireault & Godin, 2015; Amireault et al., 2015; Amireault et al., 2015).
Phase 1 and Phase 2: Change in exercise volume | 26-weeks post baseline
  The Godin Leisure Time Exercise Questionnaire will be used to measure exercise volume over 1 week. It is a self-report measure which asks respondents to give weekly frequencies and durations of strenuous, moderate, and mild aerobic activities and resistance training sessions. Together responses are summed to determine a total weekly leisure activity score. It is shown to be reliable and valid (r=.53) when classifying respondents into 'insufficiently active' and 'active' categories (Amireault & Godin, 2015; Amireault et al., 2015; Amireault et al., 2015; Godin & Shephard, 1985b). Respondents are classified as 'active' by exceeding a score of 24 on this scale (Amireault & Godin, 2015; Amireault et al., 2015; Amireault et al., 2015).

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Change in exercise volume | Baseline, 10-weeks post-baseline, 14-weeks post-baseline, 26-weeks post-baseline
  Exercise volume will also be assessed using a tracking device (Fitbit Inspire® 2 accelerometer). Adherence to Fitbit's use in cancer survivors is high [58,59] and Fitbit exercise data has demonstrated high correlation to Actigraph measures in this population [58]. Fitbit devices will be mailed to BCS at study inception and will be required to be worn for 7 consecutive days during the four primary data collections to determine their average daily and weekly minutes of MVPA and step count. BCS are not required to wear the device outside of the data collection timeframes, but can wear them if they choose.
Phase 1: Change in social support | Baseline, 10-weeks post-baseline, 14-weeks post-baseline, 26-weeks post-baseline
  A 14-item breast cancer-specific version of the Social Support Survey (SSS) will be used to assess seven dimensions of social support including: listening support, task challenge, emotional support, esteem support, reality confirmation, tangible assistance, and understanding breast cancer support. Respondents will be asked to score questions on a five-point Likert scale for each type of support rated from 1=very dissatisfied to 5=very satisfied. Higher scores represent a better outcome.
Phase 1: Change in health-related quality of life assessed by the Short-Form-12 | Baseline, 10-weeks post-baseline, 14-weeks post-baseline, 26-weeks post-baseline
  The Short-Form-12 (SF-12) will be used to assess HRQOL. The SF-12 is a self-administered questionnaire including 12 items addressing eight domains of health: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. A composite index is scaled from 0 to 100 and normalized to approximately 50 with a higher score indicating better health.
Phase 1: Change in quality of life assessed by the EuroQol-5 Dimension-3 level (EQ-5D-3L) | Baseline, 10-weeks post-baseline, 14-weeks post-baseline, 26-weeks post-baseline
  The EQ-5D-3L will also be used to assess HRQOL. The EQ-5D-3L is a two-part measure. The first part using a three-level scale (1=no problems, 2=some problems, 3=unable) to assess five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Lower scores represent better HRQOL. The second part assesses responder's perception of their health on a visual analogue scale from 0 (worst imaginable health) to 10 (best imaginable health).
Phase 1 and Phase 2: Cost of intervention arms | 10-weeks (post intervention)
  The costs of the MatchQEP program will be calculated and compared to traditional face-to face costs of QEP services. Program costs related to MatchQEP include labour, equipment, and consumables. The cost of training staff will also be excluded as staff will already be qualified for their role. Labour costs will by calculated by assessing the number of contact hours between the QEP and survivor over the 10-week program, and the unit cost of 1 hour of work by the QEP. For each 1-hour contact session, 1.5 hours of labour will be allocated to account for preparation time needed by the QEP during the phone sessions. Equipment related costs to run the MatchQEP program will include any form of device that a survivor may purchase for use at home based on the QEP recommendations (for example TheraBand or weights) and a computer and telephone for the QEP.
Phase 1: Use of health care resources | 10-weeks post-baseline, 14-weeks post-baseline, 26-weeks post-baseline
  The use of health care resources will be compared between the two groups at follow up time points using a piloted questionnaire assessing number of health care facility visits, doctor visits, procedures received, support services used, loss of work, and prescription medications used.
Phase 1 and Phase 2: Intervention adherence | 10-weeks post-baseline
  The QEP will track MatchQEP group adherence by completing a weekly session log. The QEP will record attendance of each BCS at the virtual QEP session as well as whether each individual completed the goals set from the previous session. MatchQEP group adherence is defined as the number of sessions attended divided by the total number of sessions.
  Match group adherence will be determined by the number of times the peers connect during the 10-week intervention period.
Phase 2: Resistance Exercise Self-Efficacy | Baseline, 8-weeks post-baseline, 26-weeks post-baseline
  Guide for constructing self-efficacy scales
Phase 2: Physical Self | Baseline, 8-weeks post-baseline, 26-weeks post-baseline
  Physical Self-Description Questionnaire:
Phase 2: Body Functionality appreciation | Baseline, 8-weeks post-baseline, 26-weeks post-baseline
  Functionality Appreciation Scale:

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murray RM, O'Loughlin E, Smith-Turchyn J, Fong AJ, McDonough MH, Mina DS, Arbour-Nicitopoulos KP, Trinh L, Jones JM, Bender JL, Culos-Reed SN, Tomasone JR, Vani MF, Sabiston CM. Connecting women who are diagnosed and treated for breast cancer to engage in physical activity: a two-arm randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Apr 25;17(1):96. doi: 10.1186/s13102-025-01131-4. PMID 40281585
- [Derived] Smith-Turchyn J, McCowan ME, O'Loughlin E, Fong AJ, McDonough MH, Santa Mina D, Arbour-Nicitopoulos KP, Trinh L, Jones JM, Bender JL, Culos-Reed SN, Tomasone JR, Vani MF, Sabiston CM. Connecting breast cancer survivors for exercise: protocol for a two-arm randomized controlled trial. BMC Sports Sci Med Rehabil. 2021 Oct 14;13:128. doi: 10.1186/s13102-021-00341-w. eCollection 2021. PMID 34649590
- See also: Connecting breast cancer survivors for exercise: protocol for a two-arm randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/34649590/